CLINICAL TRIAL: NCT01276210
Title: A Phase I Trial of Sorafenib and Stereotactic Radiosurgery for Patients With 1-4 Brain Metastases
Brief Title: Sorafenib Tosylate and Stereotactic Radiosurgery in Treating Patients With Brain Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, A Bapsi Chakravarthy, MD, Associate Professor; Radiation Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC RAD1060; NCI-2010-02407 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-01-11; First posted 2011-01-13 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Tumors Metastatic to Brain
MeSH Terms: conditions — Brain Neoplasms | interventions — Sorafenib; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): See Detailed Description
  Interventions: Drug: sorafenib tosylate; Radiation: stereotactic radiosurgery; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: sorafenib tosylate — Given PO
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Radiation: stereotactic radiosurgery — Undergo stereotactic radiosurgery
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
RATIONALE: Sorafenib tosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth or by blocking blood flow to the tumor. Stereotactic radiosurgery (SRS) may be able to send x-rays directly to the tumor and cause less damage to normal tissue. Giving sorafenib tosylate together with SRS may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and the best dose of sorafenib tosylate when given together with SRS in treating patients with brain metastases

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety, tolerability and maximum tolerated dose (MTD) of sorafenib, when administered in combination with SRS to patients with 1-4 metastatic brain tumors.

SECONDARY OBJECTIVES:

I. To assess the six-month intra-cranial progression-free survival (PFS) of sorafenib when administered in combination with SRS to patients with 1-4 metastatic brain tumors. PFS is defined as the time to intra-cranial tumor progression or death.

II. To assess the six-month overall survival (OS) of sorafenib when administered in combination with SRS to patients with 1-4 metastatic brain tumors.

III. To compare results to patients who are treated with SRS alone (concurrent controls).

OUTLINE: This is a dose-escalation study of sorafenib tosylate.

Patients receive oral (PO) sorafenib tosylate once daily and undergo SRS 5-7 days later. Treatment with sorafenib continues for 2 weeks after SRS in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 8, 26, and 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cancer with 1-4 brain metastases (except lymphoma or small cell histologies)
* ECOG PS 0 or 1
* Patients are candidates for stereotactic radiosurgery as determined by the treating radiation oncologist. Intra-cranial tumors must measure 4cm or less in greatest dimension. Patients may have received prior neurosurgical resection(s) of intra-cranial metastases if their operation(s) was (were) completed at least 6 months prior to study enrollment. Patients may have had prior whole brain radiation therapy (WBRT) if it was completed at least 6 months prior to study enrollment.
* Age ≥ 18 years and willing and able to sign a written informed consent; a signed informed consent must be obtained prior to any study specific procedures
* INR < 1.5 or a PT/PTT within normal limits; patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate; for patients on warfarin, the INR should be measured prior to initiation of sorafenib and monitored at least weekly (INR must be therapeutic in the range of 2-3)

Subjects must receive 1st dose of sorafenib 5-7 days prior to administration of Stereotactic Radiosurgery.

Exclusion Criteria:

* Congestive heart failure > class II NYHA; patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months
* Unable to undergo brain MRI
* CNS metastases from lymphoma or small cell lung cancer
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Uncontrolled hypertension defined as systolic blood pressure > 140mm Hg or diastolic pressure > 90 mm Hg, despite optimal medical management
* Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C
* Active clinically serious infection > CTCAE v 4.0 Grade 2
* Thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months
* Pulmonary hemorrhage/bleeding event >= CTCAE v 3.0 Grade 2 within 4 weeks of first dose of study drug
* Any other hemorrhage/bleeding event >= CTCAE v 3.0 Grade 3 within 4 weeks of first dose of study drug
* Serious non-healing wound, ulcer, or bone fracture
* Any drug that results in hepatic enzyme induction such as anti-convulsants (dilantin, depakote, tegretol, phenobarbital); keppra is allowed
* Evidence or history of bleeding diathesis or coagulopathy
* Any pulmonary hemorrhage CTCAE v 4.0 Grade 2 or higher within 4 weeks of first study drug
* Any other bleeding or hemorrhage CTCAE v 4.0 Grade 3 or higher within 4 weeks of first drug
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug
* Use of St. John's Wort or rifampin (rifampicin) within the last 8 weeks
* Known or suspected allergy to sorafenib
* Any condition that impairs patient's ability to swallow whole pills
* Concurrent investigational drugs
* Concurrent steroids are allowed if Dexamethasone dose is =< 16mg daily; if feasible, steroids should be weaned off once sorafenib has been initiated
* Prior therapy with sorafenib or other tyrosine kinase inhibitors within the last 12 months; patients are allowed to have been on prior bevacizumab therapy as long as it was stopped at least 6-8 weeks prior to enrolling on this trial
* Any malabsorption problem
* Hemoglobin =< 9.0 g/dl
* Absolute neutrophil count (ANC) =< 1,500/mm^3
* Platelet count =< 100,000/mm^3
* Total bilirubin >= 1.5 times upper limit of normal (ULN)
* ALT and AST >= 2.5 times the ULN ( =< 5 x ULN for patients with liver involvement)
* Creatinine >= 1.5 times ULN
* Women of childbearing potential with a positive serum pregnancy test performed within 7 days prior to the start of treatment; women and men of childbearing potential that do not agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation; men who do not agree to use adequate birth control for at least three months after the last administration of sorafenib
* All toxicities from prior therapies must have resolved to CTCAE v3.0 Grade I or better by the time of study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-02; Primary Completion 2015-07 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD) of combining sorafenib with SRS | At 1 month

SECONDARY OUTCOMES:
Intra-cranial progression-free survival (PFS) | At 6 months
Overall survival(OS) in study patient population | at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anuradha Chakravarthy, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/